CLINICAL TRIAL: NCT06739772
Title: Development of Implementation Toolkits to Promote HPV Self-sampling Behavior Among Women Living with HIV in Ghana
Brief Title: Development of Implementation Toolkits
Acronym: HOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Matt Asare, Assistant Professor, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21TW012728-01A1 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Self Sampling; Communication Model; Implementation Science; HIV
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPV Self sampling (Experimental): Participants in the intervention group will receive HPV self sampling and behavioral intervention
  Interventions: Behavioral: HPV Self-Sampling and Behavior Intervention; Behavioral: Participants in the intervention group will receive HPV self sampling and behavioral intervention
- Control Group (No Intervention): Participants in the control group will receive enhance standard care

INTERVENTIONS:
Behavioral: HPV Self-Sampling and Behavior Intervention — Participants in the intervention group will receive HPV self sampling and behavioral intervention
  Arms: HPV Self sampling
Behavioral: Participants in the intervention group will receive HPV self sampling and behavioral intervention — Received enhance standard care
  Arms: HPV Self sampling

SUMMARY:
The purpose of the study is to conduct an intervention program aimed at increasing HPV self-sampling among women living with HIV in Ghana.

DETAILED DESCRIPTION:
Women living with HIV, (WLWH), in low- and middle-income countries (LMICs) have a six-fold increased risk of developing cervical cancer (CC) compared to their uninfected counterparts. Our studies in Ghana show that self-sampling is acceptable, easy to use, and efficacious in detecting precancer lesions among WLWH. However, this screening mechanism has not been translated to healthcare practice in Ghana.

Systematic adaptation and implementation toolkits are needed to translate self-sampling into healthcare practices. We develop a Home-based self-collected sampling for the cervical cancer Prevention Education (HOPE) toolkits to promote cervical cancer screening in Ghana. HOPE toolkit core components such as (a) self-sample HPV testing kits and (b) the 3R (Reframe, Reprioritize, and Reform) communication model will not change as they are evidence-based. The content and the intervention delivery modalities of HOPE will go through the cultural adaptation iterative processes.

This R21 resubmission seeks to develop contextually appropriate adaptation and implementation toolkits in Ghana. A three-step approach will be used for the adaption process and evaluation of the toolkit. First, we will organize focus group discussions (FGDs) to identify contextual factors affecting the toolkit adaptation and nominal group techniques (NGTs) to determine the different compositions of the toolkits and select the final toolkit. A sample of 35 stakeholder advisory board members representing three organizational levels: potential intervention participants (i.e., WLWH), community leaders, and healthcare workers (e.g., doctors, nurses, administrators) will participate in the focus group FGDs and NGTs. Second, we will recruit 45 participants including WLWH and healthcare workers to evaluate the feasibility, acceptability, appropriateness, and adoptability of the selected toolkit. Third, we will test the preliminary efficacy of HOPE on cervical cancer screening defined as cervical cancer screening uptake among WLWH in the intervention arm (n=54) and control arm (n = 54). Participants will be recruited from the Cape Coast Teaching Hospital (CCTH). Specific aims of HOPE are:

Aim I: Develop and adapt the HOPE toolkit: Hypothesis: Stakeholders will identify and prioritize community needs and translate findings into a culturally adapted toolkit. Aim II: Evaluate the characteristics of the HOPE toolkit: Hypothesis: We hypothesize that 80% of participants will find HOPE toolkits feasible, acceptable, appropriate, and adoptable. Aim III: Assess the efficacy of HOPE on CCS. Hypothesis: We hypothesize that CCS behavior will increase significantly among women in the intervention group compared to those in the control group. Aim IV: Identify actionable factors and implementation costs that influence the adoption of the toolkit. Hypothesis: The Actionable factors and implementation costs will significantly influence the toolkit adoption.

ELIGIBILITY:
Inclusion Criteria:

* General eligibility criteria for these stakeholders include (1) the ability to give consent per Institutional Review Board stipulations, (2) residing in the central region of Ghana, (3) having no medical, psychological, or social characteristics that would interfere with the ability to fully participate, and (4) the willingness to participate in this study.

  1. Specific eligibility for Intervention participants (WLWH). Study inclusion/exclusion criteria for potential participants will be assessed using E-tracker data and include women (identified female at birth) who (1) are living with HIV between 25 and 65 years old5 and (2) have never had a cervical cancer screening like pap test or HPV test before, or have not had pap test or HPV testing for the past 5 years

Exclusion Criteria:

* Women will be excluded if they are pregnant or have had a hysterectomy. WLWH (female-identified at birth) who have a cervix are the main target population to develop the HOPE toolkit.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identified female at birth
Enrollment: 108 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Cervical cancer screening uptake | 6 weeks
  The outcome is screening uptake (i.e., the completion and return of a self-sample kit and pap test completion). Measure: The screening completion outcome will be binary (yes/no), and it will be assessed via the patient clinical records by the doctors at 6 weeks post-intervention. The screening completion outcome will be binary (yes/no)

SECONDARY OUTCOMES:
Screening Test Results | 6 weeks
  Screening test results (positive, negative, or inadequate). Measure: The screening test results (positive, negative, or inadequate), will be treated as categorical outcome and it will be assessed via the patient clinical records by the doctors at 6 weeks post-intervention.
Treatment follow-up | 6 weeks
  Whether patients with positive results follow up for treatment or not. Measures: The outcomes will be assessed via the patient clinical records by the doctors at 6 weeks post-intervention. The treatment follow-up (yes, no, or lost-to-follow-up) will be treated as categorical outcomes

OTHER OUTCOMES:
Actionable outcome : Implementation experience | 6 weeks after the intervention
  Implementation experience, including resource availability, managerial support, and technical issues confronted. Measure: Following the completion of the intervention(i.e., after 6 weeks), interviews will be conducted among healthcare providers using a semi-structured interview guide to assess the implementation experience outcome.
Actionable factor: Operational experience | 6 weeks after the intervention
  Operational experience, including workload increase or decrease, the flow of communication in the hospital, and any skills needed. Measure: Following the completion of the intervention(i.e., after 6 weeks), interviews will be conducted among healthcare providers using a semi-structured interview guide to assess the operational experience outcome.
Actionable factor: Adoption or level of endorsement | 6 weeks after the intervention
  Level of endorsement of the toolkit adoption and recommendations for maintenance. Measure: Following the completion of the intervention(i.e., after 6 weeks), interviews will be conducted among healthcare providers using a semi-structured interview guide to assess the adoption or endorsement outcome.
Implementation cost | Throughout the intervention period (about 12 months)
  Implementation costs will include (i) sampling materials, including kits and laboratory testing costs; (ii) recruitment (i.e., time spent identifying and contacting eligible women, advertising materials, participant incentives); (iii) intervention delivery; (iv) participant out-of-pocket costs (e.g., transportation, childcare, mobile data usage, time spent on the intervention); (v) clinic-based Pap tests; and (vi) treatment and biopsies. Measure: A cost-tracking database will be used throughout the study to itemize, quantify, and value the resources.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Asare, PhD, Principal Investigator — Baylor University
Locations (1):
- University of Cape Coast Teaching Hospital, Cape Coast, Central Region, Ghana

REFERENCES:
- [Derived] Asare M, Ebu Enyan NI, Sencherey VL, Lamptey-Mills E, Ken-Amoah S, Akakpo PK, Sturdivant RX, Obiri-Yeboah D. Culturally adapting and evaluating an evidence-based communication intervention with HPV self-sampling to improve cervical cancer screening among women living with HIV in Ghana: a mixed-methods study. BMJ Open. 2025 Dec 31;15(12):e105852. doi: 10.1136/bmjopen-2025-105852. PMID 41475829
- [Derived] Asare M, Obiri-Yeboah D, Ken-Amoah S, Akakpo PK, Enyan NIE, Asmah E, Sturdivant RX. HPV self-sampling for cervical cancer screening among women living with HIV in Ghana: protocol for a hybrid type 1 effectiveness-implementation randomized controlled trial. Trials. 2025 Nov 26;26(1):550. doi: 10.1186/s13063-025-09262-2. PMID 41299750